CLINICAL TRIAL: NCT07058961
Title: Study of the Intestinal Microbiota of Patients Admitted to Intensive Care for Severe Brain Injury.
Brief Title: Study of the Intestinal Microbiota
Acronym: NEUROBIOTE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0214/OB; N° IDRCB : 2023-A02007-38 (Other: ANSM)
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Intestinal Microbiota Between Different Groups
Keywords: brain-damaged patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — stool collection by rectal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients admitted to surgical intensive care
- Patients admitted to neurosurgical intensive care for serious brain injury

SUMMARY:
The intestinal microbiota is the set of numerous microorganisms (between 1012 and 1014 bacteria, viruses, parasites, and non-pathogenic fungi) that live in our digestive tract, mainly in the small intestine and colon. Like a fingerprint, the intestinal microbiota is unique to each individual. However, there is a common core of 15-20 species present in all humans, responsible for the essential functions of the microbiota.

Recent techniques for high-throughput sequencing of genetic material and metabolomics (i.e., the global analysis of the elements produced by the microbiota) have made it possible to more precisely describe the relationships between microorganisms and the host and how each influences the functioning of the body. Thus, we now know that the microbiota plays a role in digestive, metabolic, immune, and neurological functions. Certain events will modify the microbiota in a more or less lasting way: illnesses, medical treatments, diet, lifestyle. And these changes to the microbiota can, in turn, influence the body's behavior. As a result, dysbiosis-a quantitative, qualitative, or functional alteration of the microbiota-is a serious avenue for explaining certain pathologies.

This topic has become central to biological and medical research, as evidenced by the growing number of scientific publications since the 2010s. Scientists are trying to explore the bidirectional links between dysbiosis and pathologies. They are also trying to explore therapeutic avenues: how to modulate the microbiota to maintain it, bring it closer to, or restore its "normal" configuration to limit the impact of dysbiosis? Research has yielded encouraging results: fecal transplantation (instilling a sample of normal microbiota from the feces of healthy donors into a sick person) or new-generation probiotics with protective biological effects.

DETAILED DESCRIPTION:
New research data have so far failed to find concrete resonance in intensive care patients, even though this highly stressed population is subjected to harmful pressure on the microbiota: antibiotics, gastric acid inhibitors, artificial nutrition, and sedative drugs that inhibit peristalsis. Studies remain conflicting, and this lack of evidence limits the development of targeted therapies for intensive care patients. The reason lies in the fact that there is no such thing as "one" intensive care patient, but rather different profiles depending on the type and level of stress, whether or not there is a surgical insult, the route of artificial nutrition administration, and the duration of antibiotic therapy. It is therefore necessary to conduct a comprehensive assessment. This essential preliminary information will ultimately aid in the development of targeted therapies designed to restore the microbiota and hopefully improve patient prognosis. This NEUROBIOTE study is part of this research framework and aims to explore the microbiota of a homogeneous category of patients: those admitted to surgical or neurosurgical intensive care for brain injury, whether traumatic or not, and for serious brain injury (i.e., requiring intubation). During the first phase of the study, the microbiota mapping of these patients, obtained after analysis of admission stools by rectal swab, was compared with that of a "control" group: patients admitted to surgical intensive care for multiple trauma without associated brain injury or for any state of shock requiring mechanical ventilation. During the second phase, changes in the microbiota of the "brain-injured patients" group during the first week of care, in light of the evolution of various factors: nutritional support, energy metabolism using indirect calorimetry, and markers of organ failure, will be analyzed.

This pilot study will lay the groundwork for those aiming to study other specific ICU populations.

ELIGIBILITY:
Inclusion Criteria:

Brain-injured patient group: Any adult patient admitted to neurosurgical or surgical intensive care for severe brain injury, traumatic or not, requiring intubation, eligible for indirect calorimetry measurements, and whose expected length of stay is > 48 hours.

Control group: Any adult patient admitted to surgical intensive care for multiple trauma without associated brain injury and/or for shock (hemorrhagic or septic*) and whose expected length of stay is > 48 hours.

Exclusion Criteria:

* Refusal to participate in the study (request of non-opposition from relatives if the patient is unfit)
* Lack of social security affiliation;
* Minor patient;
* Patient under legal protection (guardianship or guardianship);
* Pregnant woman;
* Moribund patient or whose expected length of stay is ≤ 48 hours;
* Contraindication to indirect calorimetry (high FiO2, etc.);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient admitted to neurosurgical or surgical intensive care for severe brain injury, traumatic or not, requiring intubation, eligible for indirect calorimetry measurements, and whose expected length of stay is > 48 hours and Any adult patient admitted to surgical intensive care for multiple trauma without associated brain injury and/or for shock (hemorrhagic or septic*) and whose expected length of stay is > 48 hours.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To describe the intestinal microbiota of patients admitted to surgical or neurosurgical intensive care for severe brain injury based on analysis of admission stools by rectal swab. | At Enrollment visit and Day 28
  Analysis of the intestinal microbiota of patients admitted to surgical or neurosurgical intensive care for severe brain injury using metagenomics (composition and diversity).

SECONDARY OUTCOMES:
To compare the microbiota of patients admitted to surgical or neurosurgical intensive care for severe brain injury with that of patients with multiple trauma and/or shock. | At enrolment visit and Day 28
  Analysis of the intestinal microbiota of patients admitted to surgical intensive care for multiple trauma and/or shock requiring mechanical ventilation based on analysis of admission stools.
To analyze the changes in the intestinal microbiota of these patients as a function of nutritional interventions. | Day 7
  Analysis of the evolution of the microbiota of patients admitted to surgical intensive care for severe brain injury during the first week of hospitalization in relation to the modalities of nutritional support (calorie intake, types and routes of administration of artificial nutrition).
To analyze the changes in the intestinal microbiota of these patients as a function of anti-infectious therapies. | Day 7
  Analysis of the evolution of the microbiota of patients admitted to surgical intensive care for severe brain injury during the first week of hospitalization in relation to the modalities of anti-infectious treatment (surgical techniques and drug treatment).
To analyze the links between these modifications and the evolution of organ failures during the first week of hospitalization. | Day 7
  Evaluation of the link between evolution of the microbiota and evolution of the organ failure score (SOFA).

CONTACTS AND LOCATIONS:
Overall Officials: Emilie EO OCCHIALI, Doctor, Study Director — University Rouen Hospital
Locations (1):
- Services de Réanimation Chirurgicale Et Réanimation Neurochirurgicale, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.